CLINICAL TRIAL: NCT06169423
Title: Simulation of Perinatal Grief. Assessment of Knowledge Acquisition, Support Skills, Self-awareness and Student Satisfaction.
Brief Title: Simulation of Perinatal Grief. (SPG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JAUI_NUR_1
Record Dates: First submitted 2023-10-23; First posted 2023-12-13 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Perinatal Death; Perinatal Grief; Teaching Innovation
Keywords: Perinatal Death; Grief; Teaching Innovation; Clinical simulation
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Intervention Model Description: This is an activity for simulation-based learning.
Masking Description: The participants are nursing students. The questionnaire that they will carry out to find out their knowledge and satisfaction will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educative intervention (Other): A first theoretical session was carried out in order to acquire theoretical knowledge, skills to provide support for perinatal grief, and improve self-awareness. Prior to this, a pre-questionnaire was carried out in order to previously evaluate these aspects.
  Subsequently, a first session was held to make contact with the simulation, teach the scenarios, material, etc. This session would be the prebriefing. After this session, the complete simulation, with subsequent evaluation of it giving feedback to the students (debriefing). After this, two questionnaires were passed: one related to the acquisition of knowledge, skills to provide support, self-awareness and another on the students' satisfaction with the simulation.
  Interventions: Other: Educative intervention

INTERVENTIONS:
Other: Educative intervention — an activity for simulation-based learning First, a theoretical session was carried out in order to acquire theoretical knowledge, skills to provide support for perinatal grief, and improve self-awareness. Prior to this, a pre-questionnaire was carried out in order to previously evaluate these aspects.
  Subsequently, a first session was held to make contact with the simulation, teach the scenarios, material, etc. After this, two questionnaires were passed: one related to the acquisition of knowledge, skills to provide support, self-awareness and another on the students' satisfaction with the simulation.
  Other Names: Formative intervention

SUMMARY:
A proposal for teaching innovation is proposed with the topic of "perinatal grief" very little studied and taught in degrees such as medicine, nursing and psychology, with scientific evidence demonstrating a knowledge deficit on the part of healthcare professionals.

DETAILED DESCRIPTION:
A proposal for teaching innovation is proposed with the topic of "perinatal grief" very little studied and taught in degrees such as medicine, nursing and psychology, with scientific evidence demonstrating a knowledge deficit on the part of healthcare professionals. With the aim of improving this knowledge and the communication skills of the students who are taught, the objective is to introduce perinatal grief so that the level of knowledge on this topic increases and also increases their communication abilities in this aspect, being a very difficult topic to cover if you do not have training. To carry out teaching innovation, it is proposed, in addition to a master class to impart theoretical knowledge, to innovate by carrying out clinical simulation among students and through a questionnaire to evaluate whether this type of technique is effective for the acquisition of knowledge, skills to provide support. , improve self-awareness and also assess student satisfaction.

ELIGIBILITY:
Inclusion Criteria: The sample population will be nursing students. Specifically, the project will be proposed and offered to students who have taken the subject "Women's Care" in the third year.

-

Exclusion Criteria: Those students who did not come to class the day that the activity took place, were excluded.

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Mesure if simulation techniques are effective in helping to acquire knowledge about perinatal grief in nursing degree students. | 3 months
  Rate the knowledge acquired
Mesure if simulation techniques are effective in acquiring support skills and improving self-awareness about perinatal grief in nursing degree students. | 3 months
  Rate the effectiveness of simulation techniques
Determine the degree of satisfaction of nursing degree students with the simulation learning of how to approach perinatal grief. | 3 months
  Satisfaction questionnaire with the activity

CONTACTS AND LOCATIONS:
Locations (1):
- Isabel Almodóvar Fernández, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: Yes
If it is possible to publish in scientific journals related to the topic described, the results will be disseminated.
URL: https://doi.org/10.5281/zenodo.13137854